CLINICAL TRIAL: NCT06809452
Title: The Transdiagnostic Oncology Program (TOP): a Combined Lifestyle Intervention to Improve the Quality of Life of Cancer Survivors - a Before-and-after Pilot Study in Primary Care
Brief Title: Transdiagnostic Oncology Program in Primary Care
Acronym: TOP
Status: Completed | Type: Observational
Sponsor: Lentis Psychiatric Institute (Other)
Collaborators: Dokter Drenthe (Unknown); University Medical Center Groningen (Other); Kloosterveen, Assen (Unknown); Gezondheidscentrum Assen-Oost, Assen (Unknown)
Responsible Party: Principal Investigator, Sanne Booij, Senior researcher, Lentis Psychiatric Institute
Other Study IDs: M17.218911_TOP2
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cancer Survivor
Keywords: cancer survivor; family-doctor led aftercare program; lifestyle intervention; transdiagnostic; general practitioner; interdisciplinary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cancer survivors taking part in the program: Eligble cancer survivors who agreed to take part in TOP and in the study.
  Interventions: Behavioral: Transdiagnostic Oncologic Program
- Cancer survivors serving as controls: Eligble cancer survivors who declined to take part in TOP, but agreed to take part in the study. They serve as a convenience control group.

INTERVENTIONS:
Behavioral: Transdiagnostic Oncologic Program — The "Transdiagnostic Oncology Program" (TOP) is a 12-month interdisciplinary aftercare program aimed at improving cancer survivors' quality of life by addressing common clinical issues.
  In the first three months, participants attended two weekly 1-hour exercise sessions led by physiotherapists. Once a week, this was followed by 1-hour mind-body therapy for stress reduction. A dietitian provided an initial group session on nutrition and advised at least two personal consultations.
  Between months 3-6, exercise was reduced to once weekly, with encouragement to continue independent exercise and relaxation. A second informational session on stress and sleep hygiene was given.
  After six months, participants continued independently, meeting the family doctor quarterly to evaluate progress.
  For the participants who experienced some psychological problems, sessions with a psychologist at an institute specialized for psycho-oncology, were available.
  Groups: Cancer survivors taking part in the program

SUMMARY:
The goal of this observational study is to learn about how cancer survivors experience a relatively new 12-month interdisciplinary aftercare program called the Transdiagnostic Oncologic Program (TOP). TOP is an innovative program offered as part of routine family-doctor care among several practices in the province Drenthe, the Netherlands. It is coordinated by the family doctor and caried out by an interdisciplinary team, consisting of the family doctor, a physiotherapist, nutritionist, and optionally a psychologist. The main questions this study aims to answer are:

* Is TOP feasible and acceptable?
* Does TOP lead to improvements in quality of life in cancer survivors? Patients who were eligible for the program (n=54) were asked to participate in research as well. Everyone who participated in TOP (n=19) agreed to participate in this study as well. Those who declined participation (n=35), were asked to serve as controls, of which 16 agreed to do so.

ELIGIBILITY:
Eligibility criteria for the program and for the study were the same, with the exception that participants were willing to sign informed consent to participate in the study.

Inclusion criteria:

* being between ≥18 and ≤ 75 years old
* having been diagnosed with cancer at least 6 months ago and/or have been long-term stable.

Exclusion criteria:

* having severe physical risks due to cancer treatment and / or comorbidities
* currently undergoing intensive chemotherapy or other treatment
* having cognitive or psychosomatic complaints that interfere with successful participation
* having skin cancer, except for melanomas with metastasis
* having a life expectancy of <1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited through an e-referral program called "Zorgdomein", local papers and flyers in the waitingroom of eleven primary care clinics in Drenthe, the Netherlands. In addition, two of them (Kloosterveen and Gezondheidscentrum Assen-Oost, Assen, the Netherlands) screened their caseload for potentially eligible participants by using the International Classification of Primary Care (ICPC) code for oncology. Sixty potential participants were approached by the family doctor. The participants who were eligible and interested were called the 'intervention group' (n=19) and allocated to one of the two training locations based on where they lived. The others (n=35), who indicated no interest, were asked to serve as part of a convenience control group, called 'control group'. Sixteen of them agreed to do so. All participants agreed to participate and signed an informed consent form before starting the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Feasibility and satisfaction. | From baseline to the end of the program, after 1 year.
  Feasibility of the intervention was assessed through attrition and attendance rates and through several questions on an evaluation form at post-intervention (T2), including adverse effects. Serious adverse events were also inquired by the GP. Satisfaction with the intervention was assessed with the same evaluation form at T2.
Change in quality of life | From baseline to the end of the program, after 1 year.
  Quality of life (QoL) was measured with the validated European Organization for Research and Treatment of Cancer 30-item Quality of Life Questionnaire (EORTC QLQ-C30). From this, global health status, an overall indicator of quality of life, as well as five functioning scales (physical, emotional, cognitive, social and role) and three symptom scales (fatigue, nausea and vomiting, and pain) were used.

SECONDARY OUTCOMES:
Change in fatigue | From baseline to the end of the program, after 1 year.
  Fatigue was comprehensively assessed by the validated Dutch version of the Multidimensional Fatigue inventory (MFI); the MFI-20.
Change in mental symptoms | From baseline to the end of the program, after 1 year.
  Mental symptoms were assessed with the 21-item Depression, Anxiety and Stress Scale (DASS-21), which is a reliable and validated questionnaire.
Change in happiness | From baseline to the end of the program, after 1 year.
  Happiness, a specific aspect of quality of life, was measured with the happiness index (HI).
Change in work ability | From baseline to the end of the program, after 1 year.
  Work ability was assessed by a validated single-item question from the work ability index (WAI).
Change in work accommodations after work resumption | From baseline to the end of the program, after 1 year.
  Work accommodations after work resumption was assessed with six contextual items. Participants who resumed work at one of the assessments (T0, T1, T2) were asked to specify any work accommodations.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Gezondheidscentrum Assen-Oost, Assen, Drenthe
  - Kloosterveen, Assen, Drenthe

IPD SHARING:
Plan to Share IPD: No
The informed consent form did not include permission for sharing data with third parties. Therefore, we are legally not allowed to do so as long as the data remains pseudonymized."

REFERENCES:
- [Derived] Booij SH, Pieper A, Wester CD, Bultmann U, Waarsenburg EC, Hoenders HJR. The Transdiagnostic Oncology Program (TOP): a multidomain lifestyle intervention to improve the quality of life of cancer survivors - a before-and-after pilot study in primary care. BMC Cancer. 2025 Nov 10;25(1):1745. doi: 10.1186/s12885-025-15063-2. PMID 41214573
- See also: Information page about TOP for clients from primary care practices in Drenthe — https://www.dokterdrenthe.nl/patienten/zorg-voor-jou/top